CLINICAL TRIAL: NCT01106287
Title: A Study of Higher Single Doses of MK-0941 in Type 2 Diabetics
Brief Title: Single Doses of MK-0941 in Type 2 Diabetics (MK-0941-027)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-027; 2010_526 (Other: Merck Telerex ID Number); MK-0941-027 (Other: protocol number)
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Period 1: Placebo - Period 2: 80 mg - Period 3: 100 mg - Period 4: Placebo - Period 5: 140 mg
  Interventions: Drug: MK-0941; Drug: Comparator: Placebo
- Treatment Sequence 2 (Experimental): Period 1: 60 mg - Period 2: 80 mg - Period 3: 100 mg - Period 4: 120 mg - Period 5: Placebo
  Interventions: Drug: MK-0941; Drug: Comparator: Placebo
- Treatment Sequence 3 (Experimental): Period 1: 60 mg - Period 2: Placebo - Period 3: 100 mg - Period 4: 120 mg - Period 5: 140 mg
  Interventions: Drug: MK-0941; Drug: Comparator: Placebo
- Treatment Sequence 4 (Experimental): Period 1: 60 mg - Period 2: 80 mg - Period 3: Placebo - Period 4: 120 mg - Period 5: 140 mg
  Interventions: Drug: MK-0941; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK-0941 — A single 60, 80, 100, 120 or 140 mg oral dose of MK-0941 will be administered in each period
Drug: Comparator: Placebo — a single oral placebo will be administered in the designated period (Periods 1-5)

SUMMARY:
This study will evaluate the safety and tolerability of single doses of MK-0941 based on assessment of clinical and laboratory adverse experiences

ELIGIBILITY:
Inclusion Criteria:

* Female participants of reproductive potential must test negative for pregnancy and agree to use two acceptable methods of birth control
* Diagnosis of Type 2 Diabetes and is either being treated with diet and exercise alone or with a single or combination oral anti-hyperglycemic agent
* No treatment with three of more anti-hyperglycemic agents or any treatment regimen that includes insulin
* In good health (except for Type 2 Diabetes)
* Willingness to follow a specific diet throughout the study (consisting of 50% carbohydrates, 20%protein and 30% fat)
* Nonsmoker

Exclusion Criteria:

* History of stroke, chronic seizure or major neurological disorder
* History of cancer
* History of Type 1 Diabetes
* Recent history of eye infection
* Glaucoma or blindness
* Eye surgery (by incision or laser) within the past three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0941 60/80/100/120 mg/Pbo: Treatment Sequence 1
- MK-0941 60/80 mg/Pbo/MK-0941 120/140 mg: Treatment Sequence 2
- MK-0941 60 mg/Pbo/MK-0941 100/120/140 mg: Treatment Sequence 3
- Pbo/MK-0941 80/100 mg/Pbo/MK-0941 140 mg: Treatment Sequence 4
Period: Overall Study
Arm/Group | MK-0941 60/80/100/120 mg/Pbo | MK-0941 60/80 mg/Pbo/MK-0941 120/140 mg | MK-0941 60 mg/Pbo/MK-0941 100/120/140 mg | Pbo/MK-0941 80/100 mg/Pbo/MK-0941 140 mg
Started | 4 (One participant that discontinued the study due to a pre-treatment adverse event was replaced.) | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-0941 60/80/Pbo/ MK-0941 120/140 mg: Treatment Sequence 2
- Total: Total of all reporting groups
Arm/Group | MK-0941 60/80/100/120 mg/Pbo | MK-0941 60/80/Pbo/ MK-0941 120/140 mg | MK-0941 60 mg/Pbo/MK-0941 100/120/140 mg | Pbo/MK-0941 80/100 mg/Pbo/MK-0941 140 mg | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (7.19) | 55.0 (7.81) | 54.7 (12.10) | 52.3 (7.51) | 51.4 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 2 | 6
  Male | 4 | 1 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events During the Study
Time Frame: Up to 30 days after the last dose of study drug
Population: All participants receiving any dose of MK-0941 or placebo
Measure: Number; unit: participants
Groups:
- MK-0941 60 mg: All participants receiving a 60-mg dose of MK-0941
- MK-0941 80 mg: All participants receiving a 80-mg dose of MK-0941
- MK-0941 100 mg: All participants receiving a 100-mg dose of MK-0941
- MK-0941 120 mg: All participants receiving a 120-mg dose of MK-0941
- MK-0941 140 mg: All participants receiving a 140-mg dose of MK-0941
- Placebo: All participants receiving placebo
Arm/Group | MK-0941 60 mg | MK-0941 80 mg | MK-0941 100 mg | MK-0941 120 mg | MK-0941 140 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 9 | 13
participants
  Adverse Event | 2 | 6 | 4 | 9 | 4 | 5
  Drug-Related Adverse Event | 1 | 1 | 2 | 6 | 3 | 1

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: Only treatment-emergent adverse events were examined for this outcome measure.
Time Frame: Up to 6 weeks after the first dose of study drug
Population: All participants receiving any dose of MK-0941 of placebo.
Measure: Number; unit: participants
Arm/Group | MK-0941 60 mg | MK-0941 80 mg | MK-0941 100 mg | MK-0941 120 mg | MK-0941 140 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 9 | 13
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug
Description: The 13 study participants received multiple doses of drug at different dose levels.
Groups:
- MK-0941 60 mg: All participants receiving at least one dose of 60 mg of MK-0941
- MK-0941 80 mg: All participants receiving at least one dose of 80 mg of MK-0941
- MK-0941 100 mg: All participants receiving at least one dose of 100 mg of MK-0941
- MK-0941 120 mg: All participants receiving at least one dose of 120 mg of MK-0941
- MK-0941 140 mg: All participants receiving at least one dose of 140 mg of MK-0941
Arm/Group | MK-0941 60 mg | MK-0941 80 mg | MK-0941 100 mg | MK-0941 120 mg | MK-0941 140 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/9 | 0/9 | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 2/10 | 6/9 | 4/9 | 9/9 | 4/9 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0941 60 mg (N=10) | MK-0941 80 mg (N=9) | MK-0941 100 mg (N=9) | MK-0941 120 mg (N=9) | MK-0941 140 mg (N=9) | Placebo (N=13)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Application site irritation (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 3 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.